CLINICAL TRIAL: NCT02706210
Title: Magnetic Resonance Imaging-based Comparative Research in Different Mild Cognitive Impairment Subtype
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mudanjiang Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yang Yu, MD, Mudanjiang Medical University
Other Study IDs: MudanjiangMU
Record Dates: First submitted 2016-01-28; First posted 2016-03-11 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-03

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Diffusion Tensor Imaging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- vascular cognitive disorders pre-dementia (VCD-P)
- amnestic mild cognitive impairment (aMCI)

SUMMARY:
Dementia is one of the main chronic non-communicable diseases associated with disability, institutionalization, and mortality among elderly individuals. Alzheimer's disease (AD) and vascular dementia (VD) are considered to be the main types of dementia. A widely shared view is that future treatment strategies need to focus on treatment of the earliest stages of the disease. Mild cognitive impairment (MCI) constitutes an intermediate stage between normal aging and dementia. Vascular cognitive disorders (VCD) is an umbrella term representing a wide spectrum of cognitive disorder evoked by or associated with vascular causes. It encompasses patients suffering from a range of types of cognitive impairment, from mild impairment to VD. VCD predementia (VCD-P) is at the same stage of MCI. Amnestic MCI (aMCI) is a subtype of MCI, which is also considered to be the clinical transition stage between normal aging and AD, and has been applied to detect the emerging dementia. In VCD, infarcts or profuse white matter disease are considered the cause of cognitive decline. By contrast, AD is one of the most common progressive neurodegenerative disorders thought to be caused by amyloid aggregation and the formation of tau tangles. Both VCD-P and aMCI have a deficit in cognitive domains, and may have the same chief complaints of memory deficit. If it can be clear which will turn into what type of dementia in patients with cognitive impairment stage, it can not only make us more early intervention treatment to the patients, but also can save a lot of social resources and economic costs in clinic. By applying the resting state functional magnetic resonance (fMRI), structural magnetic resonance imaging (sMRI) and diffusion tensor magnetic resonance imaging (DTI) multimodal magnetic resonance (NMR) technology, the project comprehensive analysis comparison of neurodegenerative and blood vessels of brain function in patients with mild cognitive impairment and structural abnormalities connection mode. This project in order to reveal the cognitive impairment disease neural circuits in the development of the network connection and its change rule. People can further understand the pathogenesis of cognitive impairment, discover new will provide a scientific basis for prevention, diagnosis and treatment.

DETAILED DESCRIPTION:
The investigators use both psychological tests and neuroimage to compare the differences between the two groups.

All the participants received a battery of neuropsychological tests to assess general mental status and other cognitive domains, including visual-spatial ability, executive function, language, memory, attention, and general intellectual ability. These tests included the CDR scale, the Mini-Mental State Examination(MMSE), the Montreal Cognitive Assessment(MoCA), clock drawing test (CDT), Auditory Verbal Learning Test (AVLT), activities of daily living scale(ADL) and Hamilton Depression Scale and HIS. All these evaluations were performed by two attending neurologists.

All participants were scanned on a 3.0 T Siemens scanner within a single session.

Each participant received a magnetization prepared rapidly acquired gradient echo (MPRAGE) T1-weighted scan (repetition time [TR], 1900 ms; echo time [TE], 2.2 ms; inversion time, 900 ms; matrix, 256×256; number of excitations, 1; thickness, 1 mm; 176 slices) Resting state functional images were collected using an echo-planar imaging (EPI) sequence with the following parameters: repetition time (TR)= 2000 ms; echo time (TE)=40 ms; flip angle=90°; number of slices=28; slice thickness=4 mm; gap=1 mm; voxel size=4×4×4 mm3; and matrix=64×64. Participants were asked to lie quietly in the scanner with their eyes closed during the data acquisition. This scan lasted for 478 s. For each subject, the first five volumes were discarded to allow for T1 equilibration effects and the adaptation of the subjects to the circumstances, leaving 234 images for further analysis.

The diffusion weighted imaging scans were acquired on a 3.0T Siemens Tim Trio MRI scanner. Three diffusion echo-planar imaging sequence with one zero-weighted image (b =0 s/mm2) and thirty diffusion sensitizing orientations (b =1000 s/mm2) was used with the following specifications: slice thickness=2 mm; 90 slices; repetition time = 11000 ms; echo time = 98 ms; voxel size = 2 mm isotropic; flip angle=90°; acquisition matrix = 128 mm×116 mm .

ELIGIBILITY:
Inclusion Criteria:

* For all the participants

  1. Right-hand Chinese Han people
  2. Sufficient with Mandarin language
* For VCD-P group,

  1. Clinical diagnosis of Vascular cognitive disorders
  2. Between the stage of cognitive normal and dementia
  3. Clinical diagnosis of subcortical vascular diseases
* For aMCI group

  1. Clinical diagnosis of aMCI
  2. Between the stage of cognitive normal and dementia
  3. The hippocampal atrophy confirmed by structural MRI

Exclusion Criteria:

* psychiatric disease, neurological disorder and systemic disease
* a suffering of visual abnormalities, severe aphasia or palsy
* any medical or psychological conditions

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruited patients were outpatients who were registered at the neurology department.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
fractional anisotropy (FA) | about 3-5 years after they had a complaint of cognitive deficit
  The diffusion tensor matrix would be generated from a series of diffusion weighted images, then the three eigenvalues or diffusivities, would be calculated by matrix diagonalization. FA represents the degree of anisotropy of the diffusion of water molecules in axons and decreased FA is a frequent correlate of brain tissue injury. It is a DTI parameter without units.
axial diffusivity (AxD) | about 3-5 years after they had a complaint of cognitive deficit
  AxD represents the water diffusivity parallel to the axonal fibers, and therefore commonly linked to the microstructure of myelin. It is a DTI parameter without units.
radial diffusivity (RD) | about 3-5 years after they had a complaint of cognitive deficit
  RD components of the diffusion metric provide indices of axonal integrity, measured as longitudinal diffusivity, and myelin integrity. It is a DTI parameter without units.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Hongqi Hospital of Mudanjiang Medical Universiy, Mudanjiang, Heilongjiang, China

REFERENCES:
- [Derived] Yu Y, Zhao W, Li S, Yin C. MRI-based comparative study of different mild cognitive impairment subtypes: protocol for an observational case-control study. BMJ Open. 2017 Mar 8;7(3):e013432. doi: 10.1136/bmjopen-2016-013432. PMID 28274963